CLINICAL TRIAL: NCT06578611
Title: The Effects of Perioperative Smoking Cessation on Complications in Elderly Chinese Undergoing Spinal Fusion With Enhanced Recovery After Surgery: A Prospective Cohort Study
Brief Title: Perioperative Smoking Cessation in Elderly Chinese Undergoing Spinal Fusion
Status: Not yet recruiting | Type: Observational
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024 Elderly Spinal Fusion
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Spinal Fusion
MeSH Terms: interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Blood samples will be collected after admission for assessment of biomarkers.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-smokers: Patients who did not smoke at recruitment and during follow-up.
- Continuous smokers: Patients who smoked at recruitment and during follow-up.
  Interventions: Combination Product: Enhanced recovery after surgery
- Smoking quitters: Patients who smoked at recruitment but quitted during follow-up.
  Interventions: Combination Product: Enhanced recovery after surgery

INTERVENTIONS:
Combination Product: Enhanced recovery after surgery — Recommended pre-, intra-, and post-operative care interventions in the enhanced recovery after surgery.
  Groups: Continuous smokers; Smoking quitters

SUMMARY:
As China's society ages faster, the number of elderly patients undergoing spinal fusion surgery will gradually increase. Since elderly patients are at higher risk of postoperative complications than younger patients, minimizing complications after spinal fusion becomes a priority in postoperative rehabilitation. The purpose of this prospective cohort study is to develop an enhanced recovery after surgery program including individualized perioperative smoking cessation strategies in Chinese elderly undergoing spinal fusion.

DETAILED DESCRIPTION:
With the aging society, elderly population in China has reached 172 million (12%) in 2020 and is predicted to rise to 336 million (26%) by 2050. This will be accompanied by more elderly people with degenerative spinal diseases who may become candidates for spinal surgery (e.g., spinal fusion). Compared with younger patients, elderly patients are more likely to experience complications after spinal fusion (e.g., 9% and 14% for <65 and ≥ 65 years old in lumbar fusion), which may lead to adverse patient outcomes including worse functional outcomes and satisfaction and increased revision surgery.

Recently, enhanced recovery after surgery (ERAS) program for spinal fusion including the pre-, intra-, and post-operative care interventions has been developed. Previous studies have shown that ERAS has multiple benefits for elderly undergoing spinal fusion, such as reduced complications and shorter hospital stays. However, the preoperative smoking cessation protocols varied widely between studies (e.g., at least 4 weeks, 3 months, and 2 weeks before surgery), which may be due to a lack of evidence.

Therefore, we plan to conduct a prospective study to improve the perioperative smoking cessation strategy of ERAS and establish an evidence-derived protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 65 years old or more;
2. Patients who plan to undergo spinal fusion with ERAS program;
3. Patients who agreed to participate in this study.

Exclusion Criteria:

1. Patients who cannot understand the study content or have difficulty communicating;
2. Patients with a history of spinal fusion surgery;
3. Patients with spinal fractures, spinal tumor, or spinal infections;
4. Patients with congenital spinal deformity;
5. Patients who were unable to complete at least 6 months of follow-up;
6. Patients with incomplete clinical information.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 years old or more undergoing spinal fusion.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of any complications | From the date of surgery until 6 months after surgery or the date of death from any cause, whichever come first.
  Any major or minor complications occurs during this study will be reported.

SECONDARY OUTCOMES:
Length of hospital stay | From the date of admission until the date of discharge or the date of death from any cause, whichever come first, assessed up to 6 months.
  The period from admission to discharge will be reported.
Prevalence of postoperative pain | From the date of surgery until 6 months after surgery or the date of death from any cause, whichever come first.
  Prevalence of postoperative pain will be assessed using the numeric rating scale.
Prevalence of pain-related disability | From the date of surgery until 6 months after surgery or the date of death from any cause, whichever come first.
  Pain-related disability will be assessed using Oswestry Disability Index (ODI).
Level of quality of life | From the date of surgery until 6 months after surgery or the date of death from any cause, whichever come first.
  Quality of life after surgery will be evaluated using EuroQol-5-Dimensions-5-Level.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No